CLINICAL TRIAL: NCT01062009
Title: A Safety and Dose-escalation Study of Zinc Supplementation in Pediatric Critical Illness
Brief Title: Safety and Dose Escalation Study of Zinc Supplementation in Critically Ill Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SPID 0876
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control group (No Intervention): No intervention
- Low dose group (Active Comparator): 250 mcg/kg/day supplemental IV zinc sulfate divided every 8 hours for 7 days
  Interventions: Drug: Zinc sulfate
- Medium dose group (Active Comparator): 500 mcg/kg/day supplemental IV zinc sulfate q8 hours for 7 days
  Interventions: Drug: Zinc sulfate
- High dose group (Active Comparator): 750 mcg/kg/day supplemental IV zinc sulfate q8 hrs for 7 days
  Interventions: Drug: Zinc sulfate

INTERVENTIONS:
Drug: Zinc sulfate — Zinc sulfate 200 mcg/ml in Normal Saline
  Arms: High dose group; Low dose group; Medium dose group

SUMMARY:
The purpose of the study is 1) to determine whether administration of intravenous zinc to critically ill children is safe, and 2) to determine an appropriate dose of zinc supplementation.

DETAILED DESCRIPTION:
Our recently published studies in children with septic shock demonstrated that pediatric septic shock is characterized by large scale repression of genes that either directly depend on normal zinc homeostasis or directly participate in zinc homeostasis. Functional validation studies demonstrated that nonsurvivors of pediatric septic shock have abnormally low serum zinc concentrations. A follow-up pilot study in a general population of critically ill children demonstrated that the presence of low plasma zinc concentrations is a prevalent problem in critically ill children. In addition, low plasma zinc concentrations correlate inversely with indices of inflammation and directly with the number of organ failures. These preliminary data, coupled with the expected safety of zinc supplementation, provided the rationale for a double blinded, prospective, placebo-controlled trial of zinc supplementation in critically ill children, with the two primary study endpoints to assess efficacy being highly clinically relevant: reduction of the lymphopenia rate and improvement of glucose homeostasis. Although the proposal was well-received, the primary concern precluding funding of this trial were lack of safety and dosing data for intravenous zinc. We have therefore developed a proposal for a Phase I/II study of safety and pharmacokinetics to address these concerns. It is anticipated that data generated through this proposal will provide the necessary preliminary data to re-submit our application for an interventional efficacy trial of zinc supplementation in critically ill children

ELIGIBILITY:
Inclusion Criteria:

* Admission to pediatric intensive care unit
* Age between 1 month and 10 years
* Pediatric Risk of Mortality III score > 5, OR presence of at least 1 new organ failure
* Anticipated pediatric intensive care unit length of stay > 3 days
* Ability of parent or legal guardian to provide informed consent

Exclusion Criteria:

* Known zinc deficiency
* Pre-existing bone marrow failure
* New or existing diagnosis of diabetes mellitus
* Limitation of care orders in place
* New diagnosis of brain injury, encephalopathy
* Clinical contraindication for zinc supplementation

Ages: 30 Days to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2008-11; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Z Cvijanovich, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Childrens' Hospital & Research Center Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cvijanovich NZ, King JC, Flori HR, Gildengorin G, Wong HR. Zinc homeostasis in pediatric critical illness. Pediatr Crit Care Med. 2009 Jan;10(1):29-34. doi: 10.1097/PCC.0b013e31819371ce. PMID 19057435
- [Background] Wong HR, Shanley TP, Sakthivel B, Cvijanovich N, Lin R, Allen GL, Thomas NJ, Doctor A, Kalyanaraman M, Tofil NM, Penfil S, Monaco M, Tagavilla MA, Odoms K, Dunsmore K, Barnes M, Aronow BJ; Genomics of Pediatric SIRS/Septic Shock Investigators. Genome-level expression profiles in pediatric septic shock indicate a role for altered zinc homeostasis in poor outcome. Physiol Genomics. 2007 Jul 18;30(2):146-55. doi: 10.1152/physiolgenomics.00024.2007. Epub 2007 Mar 20. PMID 17374846

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was enrolled but withdrawn by PI due to insufficient intravenous access to obtain study labs
Period: Overall Study
Arm/Group | Control Group | Low Dose Group | Medium Dose Group | High Dose Group
Started | 7 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Low Dose Group | Medium Dose Group | High Dose Group | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 1.5 [0.6 to 4.8] | 1.8 [0.8 to 2.8] | 5.3 [1.9 to 6.4] | 2.6 [0.8 to 5.2] | 1.9 [0.65 to 5.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 3 | 14
  Male | 2 | 3 | 2 | 3 | 10
Pediatric Risk of Mortality (PRISM) III [Median (Inter-Quartile Range); unit: units on a scale] — PRISM is Pediatric Risk of Mortality score The PRISM score has 17 physiologic variables subdivided into 26 ranges. The score for each variable is summed to determine the PRISM score. The minimum score (lowest risk of mortality) is 0 and the maximum score is 70.
  units on a scale | 12 [5 to 17] | 8 [3 to 16] | 12 [6 to 19] | 9 [7 to 10] | 9 [5 to 17]
Pediatric Index of Mortality (PIM) [Median (Inter-Quartile Range); unit: percentage mortality risk] — PIM, or pediatric index of mortality, is a mortality prediction model for children in intensive care. It inputs seven variables and produces a calculated percentage mortality risk ranging from 0-100%
  percentage mortality risk | 3.4 [1.6 to 17.1] | 6.0 [4.2 to 7.2] | 7.0 [4.0 to 23.0] | 5.2 [2.8 to 7.8] | 5.9 [4 to 9.7]
Pediatric Logistic Organ Dysfunction (PELOD ) [Median (Inter-Quartile Range); unit: units on a scale] — The PeLOD (Pediatric Logistic Organ Dysfunction) score is a measure of multiple organ dysfunction that sums values for 6 organ systems (cardiovascular, respiratory, renal, hepatic, hematologic, and neurologic) to give a number between 0 and 71. The higher the number the worse the organ dysfunction and the greater the risk of mortality.
  units on a scale | 11 [4 to 11] | 11 [4 to 19] | 20 [13 to 21] | 21 [14 to 21] | 11 [2 to 21]
Number of patients with >= 2 organs failed [Number; unit: participants] | 3 | 3 | 4 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Plasma Zinc Concentration Over Time
Description: Plasma Zinc levels were measured daily during the seven day study period in each group.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Control Group | Low Dose Group | Medium Dose Group | High Dose Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/dL
  Day 1 | 51.2 (14.8) | 36.4 (8.8) | 37.7 (25.2) | 43.4 (9.7)
  Day 2 | 63.0 (10.1) | 42.1 (15.4) | 46.3 (29.1) | 71.5 (34.6)
  Day 3 | 60.3 (10.7) | 47.4 (17.8) | 52.3 (10.9) | 68.2 (33.4)
  Day 4 | 59.5 (4.3) | 54.4 (17.6) | 63.3 (18.9) | 101.9 (33.4)
  Day 5 | 57.3 (5.1) | 58.9 (12.9) | 66.8 (20.0) | 71.0 (16.9)
  Day 6 | 56.8 (7.3) | 62.6 (15.7) | 66.0 (16.8) | 114.0 (43.7)
  Day 7 | 58.7 (4.9) | 67.1 (12.2) | 67.6 (10.8) | 93.3 (8.7)

2. Primary Outcome: New Fever
Description: Because of reports of fever in patients wiht zinc overdoses, we monitored patients for new fever while on supplementation
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Control Group | Low Dose Group | Medium Dose Group | High Dose Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 0 | 2 | 1 | 0
Statistical Analysis 1: Comparison: Control Group vs Low Dose Group vs Medium Dose Group vs High Dose Group; Chi square analysis comparing number of participants with new fever in each group; Test type: Superiority or Other; p = 0.24, Chi-squared

3. Secondary Outcome: Glucose Homeostasis
Description: Patients were assigned a score based on glucose range to take into account the degree of hyperglycemia as well as the need for insulin over the course of the 7 day study period. This score is an ordinal scale ranging from 1 to 5, with a score of 1 indicating no hyperglycemia, and 5 indicating severe hyperglycemia despite insulin administration.
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control Group | Low Dose Group | Medium Dose Group | High Dose Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
units on a scale
  Day 1 | 4 [3.25 to 4] | 3.5 [3 to 4] | 4 [2.5 to 4] | 2.5 [2 to 3.75]
  Day 2 | 3.5 [2.25 to 4] | 3.5 [2.25 to 4] | 4 [4 to 4] | 2.5 [2 to 3]
  Day 3 | 3.5 [2.25 to 4] | 3.5 [2.25 to 4] | 4 [3.25 to 4] | 2 [2 to 2.75]
  Day 4 | 3 [2 to 3] | 4 [4 to 4] | 4 [4 to 4] | 2 [2 to 2.75]
  Day 5 | 3 [2 to 3] | 4 [3.25 to 4] | 4 [3.25 to 4] | 2 [2 to 3.5]
  Day 6 | 4 [2 to 4] | 3.5 [2.25 to 4] | 4 [2.5 to 4] | 3 [3 to 4]
  Day 7 | 4 [2.5 to 4] | 2.5 [2 to 3.75] | 3 [3 to 3] | 2 [1.75 to 2]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Control Group | Low Dose Group | Medium Dose Group | High Dose Group
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=6) | Low Dose Group (N=6) | Medium Dose Group (N=6) | High Dose Group (N=6)
Refractory hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — One patient developed refractory hypoxemia and had to be cannulated for extracorporeal membrane oxygenation on study day 6. He recovered and survived

LIMITATIONS AND CAVEATS:
Small sample size in each group, with multiple comparisons. The study population was varied in age and diagnosis. Plasma zinc does not reflect total body zinc status, therefore a patient with low plasma Zn may not have true zinc deficiency.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No